CLINICAL TRIAL: NCT02353832
Title: Phase II Study of Stereotactic Ablative Radiotherapy (SABR) for Low Risk Prostate Cancer With Injectable Rectal Spacer
Brief Title: Stereotactic Ablative Radiotherapy (SABR) for Low Risk Prostate Cancer With Injectable Rectal Spacer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Michael Folkert, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 092013-013
Record Dates: First submitted 2015-01-16; First posted 2015-02-03 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- No Arm (Other): Study did not have Arm(s)
  Interventions: Device: Injectable Rectal Spacer (SpaceOAR, Duraseal or equivalent)

INTERVENTIONS:
Device: Injectable Rectal Spacer (SpaceOAR, Duraseal or equivalent) — Injectable Rectal Spacer (SpaceOAR, Duraseal or equivalent PEG based product

SUMMARY:
The purpose is to determine if use of rectal spacers are effective at improving protection of rectum from high dose radiation, using rate of rectal ulceration as a surrogate measure of acute effects. It is also to determine whether it provides sufficient dosimetric benefits to warrant further clinical investigation in future SABR (Stereotactic Ablative Body Radiation) related clinical studies.

DETAILED DESCRIPTION:
A phase II study to assess safety and efficacy of the spacer injection process, ability of the spacer to effectively provide the space necessary to reduce acute events in the rectum, and also meet the SABR based rectal constraints, and to monitor stability of this process during SABR. Unlike IMRT, which uses smaller dose/fraction, when using such high dose/fraction, even a few mm of shift in spacer positioning may impact the dose that the rectum receives, and therefore, a rigorous study of stability of material during the SABR treatments will need to be determined. If there is some shift, by doing this study, we may be able to determine the margin of error that will be necessary in considering rectal organ dosimetry, based on the possible shift in positiong that may occur with the spacer over time.

As the SABR therapy is strictly local, we will select for patients with prostate cancer locally confined to the prostate gland. As such, we will select eligibility criteria of low risk patients to minimize risk of extraprostatic spread, seminal vesicle invasion, and nodal spread. Hormonal therapy may also be used to shrink prostates that are massively enlarged as this may also help further reduce length of rectum that will be irradiated. As the primary toxicity will likely be mucosal damage, we will avoid enrolling patients with pre-existing mucosal dysfunction (including those with previous radiation, TURP, very large prostate glands, inflammatory bowel disease) and immunosuppressed individuals based on our phase I experience[13]. In this way, patients will be uniformly selected in a fashion that would identify patients likely to receive benefit from the therapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be willing and capable to provide informed consent to participate in the protocol.
* Eligible patients must have appropriate staging studies identifying them as AJCC stage T1 (a, b, or c) or T2a or T2b adenocarcinoma of the prostate gland. The patient should not have direct evidence of regional or distant metastases after appropriate staging studies. Histologic confirmation of cancer will be required by biopsy performed within 180 days of registration.
* The patient's Zubrod performance status must be 0-2.
* The Gleason score should be less than or equal to 6 or 3+4 if < 50% of a 12 core biopsy was involved.
* The serum PSA should be less than or equal to 10 ng/ml.
* Study entry PSA must not be obtained during the following time frames: 10 day period following prostate biopsy; following initiation of ADT; within 30 days after discontinuation of finasteride; or within 90 days after discontinuation of dutasteride.
* Age ≥ 18 years.
* Patients may have used prior hormonal therapy, but it should be limited to no more than 9 months of therapy prior to enrollment.
* The ultrasound, or CT based volume estimation of the patient's prostate gland should be ≤ 60 grams.

Exclusion Criteria:

* Subjects who have had previous pelvic radiotherapy or have had chemotherapy or surgery for prostate cancer.
* Subjects who have plans to receive other concomitant or post treatment adjuvant antineoplastic therapy while on this protocol including surgery, cryotherapy, conventionally fractionated radiotherapy, hormonal therapy, or chemotherapy given as part of the treatment of prostate cancer.
* Subjects who have undergone previous transurethral resection of the prostate (TURP) or cryotherapy to the prostate. Subjects who have significant urinary obstructive symptoms; AUA score must be ≤15 (alpha blockers allowed).
* Subjects who have a history of significant psychiatric illness.
* Men of reproductive potential who do not agree that they or their partner will use an effective contraceptive method such as condom/diaphragm and spermacidal foam, intrauterine device (IUD), or prescription birth control pills.
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years (e.g., carcinoma in situ of the breast, oral cavity, or cervix are all permissible).
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months.
  * Transmural myocardial infarction within the last 6 months.
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration.
  * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days before registration.
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol.
  * Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients.
  * Patients with history of inflammatory colitis (including Crohn's Disease and Ulcerative colitis) are not eligible.
* Subjects with a known allergy to polyethylene glycol hydrogel (spacer material) or contraindication to spacer products (Duraseal or SpaceOAR).
* Subjects with evidence of extraprostatic extension (T3a) or seminal vesicle involvement (T3b) on clinical evaluation.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male only study
Enrollment: 44 (Actual)
Dates: Start 2014-11-06 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2021-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Folkert, MD, Principal Investigator — University of Texas Southwestern Medical Center; Michael Zelefsky, MD, Principal Investigator — Memorial Sloan Kettering Cancer Centre
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UT Southwestern Medical Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Injectable Rectal Spacer: Injectable Rectal Spacer (SpaceOAR, Duraseal or equivalent): Injectable Rectal Spacer (SpaceOAR, Duraseal or equivalent PEG based product)
Period: Overall Study
Arm/Group | Single Arm: Injectable Rectal Spacer
Started | 44
Completed | 42
Not Completed | 2
Not completed — Ineligible after enrollment | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: Injectable Rectal Spacer: Injectable Rectal Spacer (SpaceOAR, Duraseal or equivalent): Injectable Rectal Spacer (SpaceOAR, Duraseal or equivalent PEG based product
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 17
Age, Continuous [Mean (Full Range); unit: YEARS] | 70 [50 to 89]
Sex: Female, Male [Count of Participants; unit: Participants] — Male only study
  Participants
    Female | 0
    Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 8
  White | 33
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Reduction in Acute Per-prostatic Rectal Ulcer Events Events From 90%+ to <70% (Particularly in the Anterior Rectum)
Description: The effectiveness of rectal spacer use was measured to determine if they are effective at improving protection of rectum from high dose radiation, using rate of rectal ulceration as a surrogate measure of acute effects
Time Frame: Median 9 months within the end of radiation treatment
Population: Observed ulceration rate
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
percentage of participants | 13.6

2. Primary Outcome: Effectiveness of Space Creation of >= 7.5 mm in Protecting Rectum From Toxicity
Description: as for outcome 1
Time Frame: Median 9 months within the end of radiation treatment
Measure: Median (Full Range); unit: mm
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
mm | 11.5 [6.6 to 21.1]

3. Secondary Outcome: Percentage of Participants With Spacer Related Acute Toxicity
Description: Assess spacer related acute toxicity. Spacer related toxicity could be related to the procedure itself (bleeding, infection, pain), or secondary effects of spacer (erectile dysfunction, persistent pain and discomfort). Adverse events will be graded by a numerical score according to the defined NCI Common Terminology Criteria for Adverse Events (NCI CTCAE V4.0) and version number 4.0 specified in the protocol. Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe or medically significant but not immediately life threatening; Grade 4: Life threatening consequences; Grade 5: Death related to the adverse event.
Time Frame: 270 days
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
percentage of participants
  Grade I | 0
  Grade II | 0
  Grade III | 2.3
  Grade VI | 0
  Grade V | 0

4. Secondary Outcome: Determine Spacer's Ability to Change Percent Rectal Circumference (PRC) Receiving 39 Gy
Description: Determine spacer's ability to change percent rectal circumference (PRC) receiving 39 Gy by at least 50%. This will be determined by using CT planning studies for dosimetric analysis before and after spacer placement.
Time Frame: 1 month
Measure: Mean (Full Range); unit: percent rectal circumference
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 8
percent rectal circumference | 99.8 [41 to 100]

5. Secondary Outcome: Determine Spacer's Ability to Change Percent Rectal Circumference (PRC) Receiving 24 Gy.
Description: Determine spacer's ability to change percent rectal circumference (PRC) receiving 24 and 39 Gy by at least 50%. This will be determined by using CT planning studies for dosimetric analysis before and after spacer placement.
Time Frame: 1 month
Measure: Mean (Full Range); unit: percent rectal circumference
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 8
percent rectal circumference | 59.3 [24.2 to 95.9]

6. Secondary Outcome: Acute (Within 270 Days of Treatment) SABR-related Gastrointestinal (GI) Toxicities
Description: Acute gastrointestinal (GI) toxicity is defined as grade 1-5 toxicity occurring prior to 270 days from the start of protocol treatment. It is graded based on CTCAE v4.0.
Time Frame: 270 days
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
percentage of participants
  Grade I | 58.1
  Grade II | 23.3
  Grade III | 0
  Grade IV | 0
  Grade V | 0

7. Secondary Outcome: Acute (Within 270 Days of Treatment) SABR-related Genitourinary (GU) Toxicities
Description: Acute genitourinary (GU)toxicity is defined as grade 1-5 toxicity occurring prior to 270 days from the start of protocol treatment. It is graded based on CTCAE v4.0.
Time Frame: 270 days
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
percentage of participants
  Grade I | 65.1
  Grade II | 46.5
  Grade III | 2.3
  Grade IV | 0
  Grade V | 0

8. Secondary Outcome: Chronic (>270 Days From Treatment) SABR-related Genitourinary (GU) Toxicities
Description: Delayed genitourinary (GU) toxicity is defined as grade 1-5 toxicity occurring after 270 days from the start of protocol treatment. It is graded based on CTCAE v4.0. Adverse events will be graded by a numerical score according to the defined NCI Common Terminology Criteria for Adverse Events (NCI CTCAE V4.0) and version number 4.0 specified in the protocol. Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe or medically significant but not immediately life threatening; Grade 4: Life threatening consequences; Grade 5: Death related to the adverse event.
Time Frame: From day 271 up to 540 days
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 42
percentage of participants
  Grade I | 64.3
  Grade II | 33.3
  Grade III | 2.4
  Grade IV | 0
  Grade V | 0

9. Secondary Outcome: Chronic (>270 Days From Treatment) SABR-related Gastrointestinal (GI) Toxicities
Description: Delayed gastrointestinal (GI) toxicity is defined as grade 1-5 toxicity occurring after 270 days from the start of protocol treatment. It is graded based on CTCAE v4.0. Adverse events will be graded by a numerical score according to the defined NCI Common Terminology Criteria for Adverse Events (NCI CTCAE V4.0) and version number 4.0 specified in the protocol. Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe or medically significant but not immediately life threatening; Grade 4: Life threatening consequences; Grade 5: Death related to the adverse event.
Time Frame: From day 271 up to 540 days
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 42
percentage of participants
  Grade I | 33.3
  Grade II | 14.3
  Grade III | 0
  Grade IV | 0
  Grade V | 0

10. Secondary Outcome: Acute Non-GI (Gastrointestinal) and Non-GU (Genitourinary) Toxicity- Irritative
Description: Toxicity will be assessed according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 4.0.
Time Frame: 270 days
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
percentage of participants
  Grade I | 44.2
  Grade II | 37.2
  Grade III | 2.3
  Grade IV | 0
  Grade V | 0

11. Secondary Outcome: Acute Non-GI (Gastrointestinal) and Non-GU (Genitourinary) Toxicity-Obstructive
Description: Toxicity will be assessed according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 4.0.
Time Frame: 270 days
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
percentage of participants
  Grade I | 41.9
  Grade II | 11.6
  Grade III | 0
  Grade IV | 0
  Grade V | 0

12. Secondary Outcome: Acute Non-GI (Gastrointestinal) and Non-GU (Genitourinary) Toxicity-Reproductive.
Description: Toxicity will be assessed according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 4.0.
Time Frame: 270 days
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
percentage of participants
  Grade I | 32.6
  Grade II | 14.0
  Grade III | 0
  Grade IV | 0
  Grade V | 0

13. Secondary Outcome: Chronic Non-GI (Gastrointestinal) and Non-GU (Genitourinary) Toxicity-Obstructive.
Description: Toxicity will be assessed according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 4.0. Adverse events will be graded by a numerical score according to the defined NCI Common Terminology Criteria for Adverse Events (NCI CTCAE V4.0) and version number 4.0 specified in the protocol. Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe or medically significant but not immediately life threatening; Grade 4: Life threatening consequences; Grade 5: Death related to the adverse event.
Time Frame: From day 271 up to 540 days
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
percentage of participants
  Grade I | 33.3
  Grade II | 14.3
  Grade III | 2.4
  Grade IV | 0
  Grade V | 0

14. Secondary Outcome: Chronic Non-GI (Gastrointestinal) and Non-GU (Genitourinary) Toxicity-Reproductive.
Description: as for outcome 13
Time Frame: From day 271 up to 540 days
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
percentage of participants
  Grade I | 14.3
  Grade II | 14.3
  Grade III | 0
  Grade IV | 0
  Grade V | 0

15. Secondary Outcome: Chronic Non-GI (Gastrointestinal) and Non-GU (Genitourinary) Toxicity-Irritative.
Description: as for outcome 13
Time Frame: From day 271 up to 540 days
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
percentage of participants
  Grade I | 42.9
  Grade II | 28.6
  Grade III | 0
  Grade IV | 0
  Grade V | 0

16. Secondary Outcome: Freedom From Biochemical Recurrence
Description: Biochemical failure RTOG-ASTRO definition (also known as Phoenix definition) - Thus, when the PSA rises by more than 2 ng/ml above the lowest level (nadir) achieved after treatment, biochemical failure has occurred and the date of the failure is recorded at the time the nadir plus 2 ng/ml level is reached
Time Frame: 4 year
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 44
percentage of participants | 93.8

17. Secondary Outcome: Overall Survival
Description: Overall survival as measured by percentage of participants who survived at 5 years. The survival time will be measured from the date of accession to the date of death.
Time Frame: 5 year
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
percentage of participants | 95

18. Secondary Outcome: Disease-specific Survival
Description: Percentage of patients who did not die from prostate cancer at 5 years.
Time Frame: 5 year
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
percentage of participants | 100

19. Secondary Outcome: Local Relapse
Description: Percentage of patients without local relapse at 3 years. Local relapse will be measured from the date of study entry to the date of documented local relapse as determined by clinical exam.
Time Frame: 3 year
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
percentage of participants | 97.5

20. Secondary Outcome: Regional Relapse
Description: Percentage of patients without regional relapse at 3 years. Regional relapse will be measured from the date of study entry to the date of documented regional nodal recurrence or distant disease relapse.
Time Frame: 3 years
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
percentage of participants | 97.5

21. Secondary Outcome: Distant Relapse
Description: Percentage of patients without distant relapse at 3 years. Distant relapse will be measured from the date of study entry to the date of documented regional nodal recurrence or distant disease relapse.
Time Frame: 3 years
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
percentage of participants | 100

22. Secondary Outcome: EPIC (Expanded Prostate Cancer Index Composite) Bowel Function
Description: Outcomes for bowel function and effect on quality of life. Expanded Prostate Cancer Index Composite (EPIC) bowel function score (range, 0 (worst) -100 (best)). EPIC bowel urgency (percentages are for men reporting more than a small problem). EPIC bowel frequency (percentages are for men reporting more than a small problem). EPIC bowel leakage or fecal incontinence (percentages are for men having fecal incontinence at least once per week). EPIC bloody stools (percentages are for men having bloody stools half the time or more). EPIC bowel, pelvic, or rectal pain (percentages are for men reporting more than a small problem). EPIC bowel habits (percentages are for men reporting more than a small problem).
Time Frame: 18 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
score on a scale | 92 [0 to 100]

23. Secondary Outcome: EPIC (Expanded Prostate Cancer Index Composite) Bowel Frequency
Description: Outcomes for bowel function and effect on quality of life. Expanded Prostate Cancer Index Composite (EPIC) bowel function score (range, 0-100). EPIC bowel urgency (percentages are for men reporting more than a small problem). EPIC bowel frequency (percentages are for men reporting more than a small problem). EPIC bowel leakage or fecal incontinence (percentages are for men having fecal incontinence at least once per week). EPIC bloody stools (percentages are for men having bloody stools half the time or more). EPIC bowel, pelvic, or rectal pain (percentages are for men reporting more than a small problem). EPIC bowel habits (percentages are for men reporting more than a small problem).
Time Frame: 18 months
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
percentage of participants | 8.25

24. Secondary Outcome: EPIC (Expanded Prostate Cancer Index Composite) Bloody Stools
Description: as for outcome 23
Time Frame: 18 months
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
percentage of participants | 0

25. Secondary Outcome: EPIC (Expanded Prostate Cancer Index Composite) Bowel Habits
Description: as for outcome 23
Time Frame: 18 months
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
percentage of participants | 25

26. Secondary Outcome: EPIC (Expanded Prostate Cancer Index Composite) Bowel Urgency
Description: as for outcome 23
Time Frame: 18 months
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
percentage of participants | 12.38

27. Secondary Outcome: EPIC (Expanded Prostate Cancer Index Composite) Bowel Leakage/Fecal Incontinence
Description: as for outcome 23
Time Frame: 18 months
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
percentage of participants | 4.125

28. Secondary Outcome: EPIC (Expanded Prostate Cancer Index Composite) Bowel Pelvic/Rectal Pain
Description: as for outcome 23
Time Frame: 18 months
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
percentage of participants | 5

29. Secondary Outcome: EPIC (Expanded Prostate Cancer Index Composite) Urinary Function
Description: Outcomes for urinary function and effect on quality of life. Expanded Prostate Cancer Index Composite (EPIC) urinary function score (range, 0 (worst)-100 (best)). EPIC urinary irritation or obstruction (range, 0-100).EPIC urinary incontinence (range, 0-100).
Time Frame: 18 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
score on a scale | 90 [0 to 100]

30. Secondary Outcome: EPIC (Expanded Prostate Cancer Index Composite) Urinary Irritative/Obstructive
Description: Outcomes for urinary function and effect on quality of life. Expanded Prostate Cancer Index Composite (EPIC) urinary function score (range, 0-100). EPIC urinary irritation or obstruction (range, 0 (worst)-100 (best)).EPIC urinary incontinence (range, 0-100).
Time Frame: 18 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
score on a scale | 88 [0 to 100]

31. Secondary Outcome: EPIC (Expanded Prostate Cancer Index Composite) Urinary Incontinence
Description: Outcomes for urinary function and effect on quality of life. Expanded Prostate Cancer Index Composite (EPIC) urinary function score (range, 0-100). EPIC urinary irritation or obstruction (range, 0-100).EPIC urinary incontinence (range, 0 (worst)-100 (best)).
Time Frame: 18 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
score on a scale | 84 [0 to 100]

32. Secondary Outcome: AUA (American Urological Association) Quality of Life Questionnaire
Description: AUA Questionnaire is used to measure urinary symptoms. AUA uses a 7-item self-report measure used to assess urinary urgency, frequency, and voiding symptoms. SYMPTOM SCORE: 0-7 (Mild) 8-19 (Moderate) 20-35 (Severe)
Time Frame: 18 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Single Arm: Injectable Rectal Spacer
Number analyzed (Participants) | 43
score on a scale | 8 [4 to 12]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality assessed for up to 5 years. Serious and Other Adverse Events assessed for up to 540 days.
Arm/Group | Single Arm: Injectable Rectal Spacer
All-Cause Mortality (participants affected / at risk) | 2/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 20/44
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm: Injectable Rectal Spacer (N=44)
Abdominal Pain (Gastrointestinal disorders) | 2
Anal Pain (Gastrointestinal disorders) | 5
Anorexia (Gastrointestinal disorders) | 10 — Loss of Appetite
Constipation (Gastrointestinal disorders) | 13
Diarrhea (Gastrointestinal disorders) | 10
Fecal Incontinence (Gastrointestinal disorders) | 4
Flatulence (Gastrointestinal disorders) | 10
Bowel Frequency (Gastrointestinal disorders) | 10
Bowel Urgency (Gastrointestinal disorders) | 7
Tenesmus (Gastrointestinal disorders) | 10
Gastrointestinal Pain (Gastrointestinal disorders) | 10
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 10
Hemorrhoids (Gastrointestinal disorders) | 4
Pelvic Pain (Gastrointestinal disorders) | 10
Perineal Pain (Gastrointestinal disorders) | 10
Proctitis (Gastrointestinal disorders) | 16
Rectal Hemorrhage (Gastrointestinal disorders) | 10
Rectal Pain (Gastrointestinal disorders) | 13
Rectal Ulcer (Gastrointestinal disorders) | 7
Telangiectasia (Gastrointestinal disorders) | 10
Bladder Spasm (Renal and urinary disorders) | 10 — Non-Sexual Domain
Cystitis Noninfective (Renal and urinary disorders) | 8 — Non-Sexual Domain
Genital Edema (Renal and urinary disorders) | 10 — Non-Sexual Domain
Hematuria (Renal and urinary disorders) | 4 — Non-Sexual Domain
Infection, Site of Spacer (Renal and urinary disorders) | 14 — Non-Sexual Domain
Prostatic Infection (Renal and urinary disorders) | 2 — Non-Sexual Domain
Prostatic Obstruction (Renal and urinary disorders) | 2 — Non-Sexual Domain
Dysuria (Renal and urinary disorders) | 10 — Non-Sexual Domain
Urinary Tract Infection (Renal and urinary disorders) | 10 — Non-Sexual Domain
Weak Urine Stream (Renal and urinary disorders) | 15 — Non-Sexual Domain
Scrotal Pain (Renal and urinary disorders) | 10 — Non-Sexual Domain
Urinary Frequency (Renal and urinary disorders) | 10 — Non-Sexual Domain
Urinary Incontinence (Renal and urinary disorders) | 14 — Non-Sexual Domain
Urinary Obstruction (Renal and urinary disorders) | 2 — Non-Sexual Domain
Urinary Retention (Renal and urinary disorders) | 13 — Non-Sexual Domain
Urinary Tract Pain (Renal and urinary disorders) | 3 — Non-Sexual Domain
Urinary Urgency (Renal and urinary disorders) | 14 — Non-Sexual Domain
Decreased Libido (Renal and urinary disorders) | 3 — Sexual Domain
Ejaculation Disorder (Reproductive system and breast disorders) | 5 — Sexual Domain
Erectile Dysfunction (Reproductive system and breast disorders) | 4 — Sexual Domain
Blood in Semen (Reproductive system and breast disorders) | 10 — Sexual Domain
Anxiety (General disorders) | 10
Fatigue (General disorders) | 7
Fever (General disorders) | 10
Paresthesia (General disorders) | 10
Rash Acneiform (Skin and subcutaneous tissue disorders) | 10
Weight Gain (General disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/32/NCT02353832/Prot_SAP_001.pdf